CLINICAL TRIAL: NCT05069441
Title: The First Affiliated Hospital of Chongqing Medical University
Brief Title: Prediction of Extubation Failure: A Multicenter Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, Principal Investigator, Chongqing Medical University
Other Study IDs: ChongqingMU4
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Mechanical Ventilation
Keywords: Extubation Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with extubation after a weaning trial: Patients who sucessfully complete a spontaneous breathing trial are enrolled in this group.

SUMMARY:
The investigators intend to collect several variables to predict extubation failure among patients who successfully complete a spontaneous breathing trial, and then develop a scale using simple bedside indicators to predict extubation failure.

DETAILED DESCRIPTION:
Mechanically ventilated patients who successfully completed a spontaneous breathing trial and prepared for extubation are eligible to enroll in this study. The vital signs, arterial blood gas tests, cough strength, cuff leak test, use of noninvasive ventilation et al. are collected. Patients are followed up to postextubation 28-day or discharge. Extubation failure is defined as reintubatin or death within postextubation 7 days. First, we will analyze the data to predict extubation failure. Then, we will combine several easily obtained variables to develop and validate a scale to predict extubation failure. Finally, we explore the predictive power of extubation failure tested by the scale and find the cutoff value to distinguish the low, moderate and high risk of extubation failure.

ELIGIBILITY:
Inclusion Criteria:

* Prepared for extubation through spontaneous breathing trial;Oral or nasal endotracheal intubation; be at least 18 years old

Exclusion Criteria:

* Extubation without a spontaneous breathing trial ;Reintubation due to secondary surgery; Tracheotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is that the patients who passed a spontaneous breathing trial and readiness for extubation.
Sampling Method: Non-Probability Sample
Enrollment: 2604 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of extubation failure | From extubation to 48 hours
  Extubation failure was defined as the reintubation or death
Rate of extubation failure | From extubation to 7 days
  Extubation failure was defined as the reintubation or death
Rate of extubation failure | From extubation to 28 days
  Extubation failure was defined as the reintubation or death

SECONDARY OUTCOMES:
Rate of mortality | From extubation to 28 days
  Mortality in ICU and hospital
ICU stay | From extubation to 28 days
  Length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jun Duan, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China